CLINICAL TRIAL: NCT02169648
Title: Study on the Correlation Between the Treatment Effectiveness of Ranibizumab and the Role of the Cytokines in Macular Edema With Retinal Vein Occlusion
Brief Title: Development of Intravitreal Ranibizumab by Determining the Pathogenesis of Macular Edema With Retinal Vein Occlusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tokyo Medical University (Other)
Responsible Party: Principal Investigator, Hidetaka Noma, Department of Ophthalmology, Hachioji Medical Center, Tokyo Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-4
Record Dates: First submitted 2014-06-13; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Macular Edema; Branch Retinal Vein Occlusion; Central Retinal Vein Occlusion
Keywords: macular edema; branch retinal vein occlusion; central retinal vein occlusion; ranibizumab; cytokines; visual acuity; central macular thickness
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ranibizumab (Experimental): Experimental: Intravitreal injection of Ranibizumab
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — intravitreal injection of 0.50 mg (0.05ml) ranibizumab monthly as needed.
  Other Names: Lucentis

SUMMARY:
The purpose of this study is to evaluate the efficacy of intravitreal ranibizumab by determining the pathogenesis of macular edema, which cause a direct effect on visual function. In particular, we focus on the correlation between the treatment effectiveness of ranibizumab and the role of the cytokines involved in the cause of macular edema.

DETAILED DESCRIPTION:
Methodology:

Aqueous humor samples (0.1ml) were obtained during intravitreous injection of ranibizumab to measure the levels of cytokines. Targeted cytokines are follows; IL-1, IL-2, IL-6, IL-8, IL-9, IL-10, IL-12, IL-13, IP-10, MCP-1, MMP-1, MIP-1β, PDGF, VEGF, PlGF, ICAM-1, TNF-α, RANTES, VEGFR-1, VEGFR-2, which has been reported that the expression level is increased in macular edema associated with RVO. Cytokines are measured by multiple ELISA (Luminex). Aqueous humor samples are obtained in the same manner from patients recurred after the first injection or continuous monthly injections. Statistical analysis is conducted to examine the difference of cytokine levels between early or late/incomplete responders of ranibizumab, and predict the number of injections to stabilize cytokine levels.

Number of centers & patients: Single center, 100 patients

Sample size justification: Sample size calculation was not done, since this study is a single-arm, observational study.

Population: Inclusion criteria: patients with RVO and macular edema

ELIGIBILITY:
Inclusion Criteria:

* Foveal thickness > 300 μm
* Best corrected visual acuity < 20/30

Exclusion Criteria:

* History of retinal diseases other than BRVO, glaucoma, uveitis, diabetes mellitus, rubeosis iridis, ocular infections, laser photocoagulation, and intraocular surgery

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Visual function by ranibizumab in macular edema with retnal vein occlusion | one year
  Mean change in central retinal thickness (CRT) and best corrected visual acuity (BCVA) at month 12

SECONDARY OUTCOMES:
Cytokine levels by ranibizumab in macular edema with retnal vein occlusion | one year
  1. Correlation between cytokine levels and mean change in CRT and/or BCVA at month 3, 6, 12,
  2. Correlation between cytokine levels and number of ranibizumab injections at month 6, 12

CONTACTS AND LOCATIONS:
Overall Officials: Hidetaka Noma, MD, Principal Investigator — Hachioji Medical Center, Tokyo Medical University
Locations (1):
- Hachioji Medical Center, Tokyo Medical University, Tokyo, Japan